CLINICAL TRIAL: NCT06276504
Title: Pembrolizumab in Progressive Multifocal Leukoencephalopathy (PML) in Immunocompromised Patients Without HIV Infection
Acronym: PENALTY
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP211001; 2023-503520-31-00 (Other: EU CT number)
Record Dates: First submitted 2024-02-14; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: Progressive Multifocal Leukoencephalopathy; Checkpoint inhibitors; Pembrolizumab
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal | interventions — pembrolizumab; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab (commercial name: KEYTRUDA; MSD), 25 mg/ml solution for intravenous (IV) injection
  Interventions: Drug: Pembrolizumab, 25 mg/ml solution for intravenous (IV) injection

INTERVENTIONS:
Drug: Pembrolizumab, 25 mg/ml solution for intravenous (IV) injection — Pembrolizumab administration at D0, M1 and M2

SUMMARY:
This study aims to assess the efficacy and safety of pembrolizumab in immunocompromised patients with progressive multifocal leukoencephalopathy (PML). This phase II, multicenter, single-arm study includes patients with an underlying cause of immunosuppression hardly reversible, i.e. not the patients with HIV nor those receiving biologics for chronic inflammatory diseases. Patients will receive intravenous pembrolizumab (2 mg/kg, maximum 200 mg) at month 0, 1 and 2 (total of three doses). The primary endpoint will be achieving at least one negative result of JCV viral load in cerebrospinal fluid (CSF) within the M0 to M3 period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Diagnosis of definite PML since less than 2 months according to American Academy of Neurology
3. Presence of JCV in the CSF in the last CSF sampling.
4. Signed informed consent (from the patient, or if unable to consent, from a surrogate)
5. For women of childbearing potential: negative serum or urine b-HCG test and agree to use a highly effective contraception methods during 8 months (i.e. until 6 months after end of experimental treatment)

Exclusion Criteria:

1. Patients in whom immune reconstitution is achievable (HIV infection - Multiple sclerosis - Auto-immune and inflammatory diseases)
2. Patients who have received solid organ transplantation
3. Hypersensitivity to the active substance or to any of the excipients
4. Life expectancy less than 1 month
5. Pregnancy or lactating women or planning birth during the study period
6. Having previously been treated by anti-PD1mAb
7. Patient receiving IL-2 or IL-7 for the treatment of PML at inclusion
8. Patient whose weight is > 100kg
9. Participation in other interventional study [a patient already included in another interventional study for which the treatment can lead to an immunodepression can be included if:

   * the investigational treatment has been completed and there is no risk of drug interaction with the administration of Pembrolizumab as defined in PENALTY study
   * if this does not alter the study's ability to evaluate the effect of Pembrolizumab in terms of safety and efficacy (from the investigator's point of view)]
10. Patient without national health insurance, and patient on AME (state medical aid)
11. Patient under guardianship or curatorship
12. Patient deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Negativation of JCV viral load in the CSF as assessed by PCR: at least one JCV PCR in the CSF negative in the Day 0 to Month 3 period | At baseline (Day 0), 1 month, 2 months and 3 months

SECONDARY OUTCOMES:
Negativation of JCV PCR viral load in the CSF: cumulative incidence of negative JCV viral load measures by PCR in CSF, with death as competing event | At baseline (Day 0), 1 month, 2 months and 3 months
Evolution of the JCV viral load in the CSF (repeated measures JCV PCR in CSF) | At baseline (Day 0), 1 month, 2 months and 3 months
Repositivation of JCV PCR: at least a positive result following at least a negative result | At baseline (Day 0), 1 month, 2 months and 3 months
Evolution of National Institutes of Health Stroke Scale (NIHSS) score | At baseline (Day 0), 1 month, 2 months, 3 months, 6 months, and 12 months
  Repeated measures of neurological status
Evolution of 6-item Modified Rankin Scale score (includes death as most severe state) | At baseline (Day 0), 1 month, 2 months, 3 months, 6 months, and 12 months
  Repeated measures of degree of disability or dependence in the daily activities in neurological conditions
Evolution of Glasgow Outcome Scale Extended (GOS-E) score | At baseline (Day 0), 1 month, 2 months, 3 months, 6 months, and 12 months
  Repeated measures of neurological outcome and degree of disability in neurological conditions
Relapse or progression | From baseline to end of participation, a maximum of 12 months
  Adjudication by a dedicated committee ; based on clinical evolution, JCV PCR in CSF, brain MRI
Death (and date of death) | From baseline to end of participation, a maximum of 12 months
Cause specific death: death related to PML | From baseline to end of participation, a maximum of 12 months
  Adjudication by a dedicated committee
Any adverse event classified by using US NCI CTCAE | From baseline to end of participation, a maximum of 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Pitié-Salpêtrière - Médecine Intensive Réanimation, Paris
  - Hôpital Pitié-Salpêtrière - Service d'hématologie clinique, Paris
  - Hôpital Pitié-Salpêtrière - Service des Maladies infectieuses et tropicales, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.